CLINICAL TRIAL: NCT07083726
Title: Smart Steps to Growth: Unleashing AI for Assessing Motor Skills in School Children
Status: Active, not recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202401852B0
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-07

CONDITIONS: AIMAS; Developmental Coordination Disorder
Keywords: Schoolchildren; Assessment; Artificial Intelligence; Motor; Developmental coordination disorder
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Samples with DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Typically Developing Children: School-age children aged 6 to 12 years who do not have a diagnosis of developmental coordination disorder (DCD).
- Developmental Coordination Disorder children: School-age children aged 6 to 12 years who have a confirmed diagnosis of DCD.

SUMMARY:
The purpose of this study is to develop an AI-based automated motor function assessment system (AIMAS) to improve early identification of developmental coordination disorder (DCD) in school-age children. The main hypothesis for this study is: Integrating AI into motor skill assessments will enhance the reliability, validity, efficiency, and accuracy of evaluating motor performance in children aged 6 to 12.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years.
* For DCD group: formal diagnosis of Developmental Coordination Disorder (DCD).
* For typically developing group: no disabilities or developmental delays.

Exclusion Criteria:

* Acute illnesses (e.g., pneumonia, upper gastrointestinal hemorrhage).
* Significant developmental delays or disabilities.
* Genetic diseases or disorders.
* Neurological disorders or injuries.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will recruit 250 school-age children, aged 6 to 12, including 170 typically developing children and 80 children with DCD.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Motor Function Assessment Score | Baseline
  AI-based Motor Function Test (Higher scores indicate better motor performance and lower risk of Developmental Coordination Disorder (DCD).)
DCD Risk Classification | Baseline
  AIMAS System Classification (System's ability to identify children at risk of DCD, compared to clinical diagnosis.)

SECONDARY OUTCOMES:
The Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan